CLINICAL TRIAL: NCT03313765
Title: A Brief Motivational Interviewing-based Intervention to Improve HIV Pre-exposure Prophylaxis Uptake Among Men Who Have Sex With Men
Brief Title: MI-based PrEP Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34DA042648 (NIH)
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2019-03

CONDITIONS: PrEP Uptake
MeSH Terms: interventions — Motivational Interviewing; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Motivational interviewing (MI)
- Standard-of-care (Active Comparator)
  Interventions: Other: Standard-of-care

INTERVENTIONS:
Behavioral: Motivational interviewing (MI) — Brief MI intervention
  Arms: Intervention
Other: Standard-of-care — Standard-of-care education and counseling
  Arms: Standard-of-care

SUMMARY:
Gay, bisexual and other men who have sex with men (MSM) are the group at highest risk of HIV infection in the United States. Pre-exposure prophylaxis (PrEP) has demonstrated high efficacy in preventing HIV infection among MSM. However, uptake in clinical settings has been slow for several reasons, including low awareness and education, low perceived HIV risk, concern for side-effects, and stigma associated with taking the medication. The purpose of the proposed study is to develop and evaluate a brief motivational interviewing (MI) intervention to promote PrEP uptake among MSM during the course of routine HIV screening at a public sexually transmitted disease (STD) clinic.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Assigned male at birth and currently identify as male
3. Score at least 10 on the HIV Incident Risk Index for MSM
4. HIV-negative based on results of antibody test
5. English- or Spanish-speaking
6. Have access to a working phone
7. Have not taken PrEP

Exclusion Criteria:

1. Have previously taken PrEP
2. Symptoms of acute HIV infection at baseline
3. HIV positive
4. A clinical contraindication to PrEP (e.g., renal dysfunction)
5. Non-English or non-Spanish speaking

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Enrollment of men who have sex with men (MSM) only
Enrollment: 86 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
PrEP uptake | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Chan, MD, Principal Investigator — Brown University/The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No